CLINICAL TRIAL: NCT02435862
Title: Protocol PVD-202: A Phase 2, Randomized, Double-Masked, Placebo-Controlled Multicenter Clinical Trial Designed to Evaluate the Safety and Efficacy Study of Luminate® in Inducing PVD in Non-Proliferative Diabetic Retinopathy
Brief Title: A Clinical Trial Designed to Evaluate the Safety and Efficacy Study of Luminate® in Inducing PVD (Posterior Vitreous Detachment) in Non-Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allegro Ophthalmics, LLC (Industry)
Collaborators: Duke University (Other); Trial Runners, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PVD-202
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Non-Proliferative Diabetic Retinopathy
Keywords: Vitreolysis of the Vitreous
MeSH Terms: interventions — risuteganib; Intravitreal Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1.0mg Luminate® (Experimental): 1.0mg Luminate® injections at day 0, 30, and 60 (day 30 and 60 if a stage 4 PVD is not present)
  Interventions: Drug: 1.0mg Luminate®
- 2.0mg Luminate® (Experimental): 2.0mg Luminate® injections at day 0, 30, and 60 (day 30 and 60 if a stage 4 PVD is not present)
  Interventions: Drug: 2.0mg Luminate®
- 3.0mg Luminate® (Experimental): 3.0mg Luminate® injections at day 0, 30, and 60 (day 30 and 60 if a stage 4 PVD is not present)
  Interventions: Drug: 3.0mg Luminate®
- Balanced Salt Solution 0.10cc (Placebo Comparator): Balanced Salt Solution 0.10cc injections at day 0, 30, and 60 (day 30 and 60 if a stage 4 PVD is not present)
  Interventions: Other: Balanced Salt Solution for intravitreal injection in 0.10cc

INTERVENTIONS:
Drug: 1.0mg Luminate®
  Arms: 1.0mg Luminate®
Drug: 2.0mg Luminate®
  Arms: 2.0mg Luminate®
Drug: 3.0mg Luminate®
  Arms: 3.0mg Luminate®
Other: Balanced Salt Solution for intravitreal injection in 0.10cc
  Arms: Balanced Salt Solution 0.10cc

SUMMARY:
A Phase 2, Randomized, Double-masked, Placebo-controlled Multicenter Clinical Trial Designed to Evaluate the Safety and Efficacy of Luminate in Inducing PVD in Subjects with Non-Proliferative Diabetic Retinopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Non-Proliferative Diabetic Retinopathy Subjects of any grade
2. Subjects with either a) no PVD, b) stage 1 PVD or c) stage 2 PVD at baseline by b-scan in the study eye
3. Subjects that are at least 45 years of age
4. Subjects that are free of other significant retinal pathologies that could interfere with the measurements or conduct of this study
5. Intraocular Pressure under control, IOP 30 mm or less
6. Male or female subjects
7. Signed Informed Consent -

Exclusion Criteria:

1. No media opacities or abnormalities that would preclude observation of the retina or performance of any study related imaging tests
2. History of prior vitrectomy in the study eye
3. Subjects with epiretinal membranes, vitreomacular adhesion, vitreomacular traction, or macular holes in the study eye at baseline
4. Subjects with proliferative DR, neovascular AMD, or retinal vascular occlusion in the study eye
5. Subjects with clinically significant macular edema in the study eye
6. Subjects with a history of focal/grid or pan-retinal laser photocoagulation in the study eye
7. Subjects likely to need intraocular surgery, laser treatment, or non-study intravitreal injections in the study eye during the study period.
8. Subjects with history of retinal detachment in the study eye
9. High myopes with a spherical equivalent of > -8.00 D spectacle correction in the study eye
10. Subjects with systolic BP> 180 at screening
11. Subjects with HgA1c >12.0 within 90 days preceding enrollment
12. Subjects that have chronic or recurrent uveitis
13. Subjects that have ongoing ocular infection or inflammation
14. Subjects with uncontrolled glaucoma, ie IOP > 25mm with or without IOP lowering agents
15. Subjects that have contraindications to the study medication
16. Subjects who are unable to meet the extensive post-op evaluation regimen
17. Pregnant or nursing women
18. Subjects with a history of penetrating ocular trauma in the study eye
19. Subjects that are participating in another clinical research study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Observation of pharmacologic induction of PVD. | 90 days
  The primary endpoint of this study is observation of pharmacologic induction of at least a stage 3 PVD, with PVD defined as a complete PVD to the equator except for vitreopapillary adhesion as seen on B-scan Ultrasound and confirmed by OCT where possible by study day 90 as determined by the reading center.

SECONDARY OUTCOMES:
The secondary endpoints of this study is the observation of a complete stage 4 PVD to the equator including vitreopapillary release as seen by B-scan ultrasound and confirmed by OCT where possible by study day 90 as determined by the reading center. | 90 days
  The secondary endpoints of this study is the observation of a complete stage 4 PVD to the equator including vitreopapillary release as seen by B-scan ultrasound and confirmed by OCT where possible by study day 90 as determined by the reading center.

CONTACTS AND LOCATIONS:
Overall Officials: Vicken Karageozian, MD, Study Director — Medical monitor
Locations (12):
- United States (12):
  - Northern California Retina Vitreous Associates, Mountain View, California
  - UCI Medical Center, Orange, California
  - New England Retina Associates, New London, Connecticut
  - Center for Retina and Macular Disease, Lakeland, Florida
  - Illinois Retina Center, Springfield, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Retina Research Institute Of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Valley Retina Institute, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - The Retina Group of Washington, Fairfax, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington